CLINICAL TRIAL: NCT04281212
Title: Prospective, Multicentric Observational Study Evaluating the Management of Chronic Coronary Occlusions In France
Brief Title: Observational Study Evaluating the Management of Chronic Coronary Occlusions In France
Acronym: ENCOCHE
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 19.05.21.62908; 2019-A01395-52 (Other: ANSM, France)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Coronary Occlusion
Keywords: Chronic Coronary Occlusion; Peripheral Component Interconnect; Coronary angioplasty
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTO: Period of 1 month in the participating centers, during which all the patients with CTO and responding to all selection criteria may be included in the study, in order to describe which therapeutic choices have been chosen for this type of patient.
- CTO with attempted angioplasty: Period of 2 months in the participating centers, during which all the patients for whom an angioplasty has been attempted after a CTO, and responding to all selection criteria, may be included in the study, in order to evaluate the success of the procedure

SUMMARY:
Data from the literature on the management of Chronic Coronary Occlusions (CTO) in France highlight a lack of epidemiological data on these patients at the national level.

For this reason, it was decided to set up this large-scale survey in order to have a picture of the management of patients with chronic coronary occlusion in France, to study the prevalence of CTOs in France as well as their management (medical, surgical or interventional), and then by analysing more precisely, over a second survey period, CTO angioplasties in terms of success rates, complications, medico-economic impact.

DETAILED DESCRIPTION:
This exhaustive and descriptive study of CTO patients, performed on a set of approximately 100 interventional cardiology centers in France, will be conducted in two steps:

* 1st step: This collection will be done over one month, the objective of which will be to photograph the therapeutic choice in the management of CTO (drug, surgical, endovascular approach).
* 2nd step: a second collection will be carried out over a period of two months, the objective of which will be to evaluate, in patients presenting a CTO with an attempt at angioplasty, the success of the procedure.

ELIGIBILITY:
Phase I

Inclusion Criteria:

* Patient over 18 years old
* Patient with CTO

Exclusion Criteria:

* Patient with acute occlusion or subocclusive lesion or CTO of less than 3 months
* Patient expressing his refusal to participate in the observatory

Phase II

Inclusion Criteria:

* Patient over 18 years old
* Patient with CTO who has attempted angioplasty

Exclusion Criteria:

* Patient with acute occlusion or less than 3 months.
* Patient demonstrating refusal to participate in the observatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As defined by the European CTO Club consensus, a chronic occlusion (CTO) is a total coronary occlusion, TIMI 0 (without anterograde coronary flow), more than 3 months old.
  To assess the CTO, the JCTO score will be used to assess the clinical and angiographic criteria of the lesions.
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Choice of treatment in management of patients with CTO | Through the end of hospitalization, an average of 5 days
  Rate of patients with CTO treated by medical treatment alone and/or by surgery, and/or by angioplasty
Success of the angioplasty for management of CTO | Through the end of hospitalization, an average of 5 days
  Procedural success rate defined by residual stenosis ≤ 30% with a TIMI (Thrombolysis In Myocardial Infarction) 3 flow and no hospital complications at the end of the angioplasty procedure

SECONDARY OUTCOMES:
Rate of events occured after procedure of angioplasty during the hospitalization, for patients with CTO | Through the end of hospitalization, an average of 5 days
  Major Adverse Cardiac and Cerebrovascular Events (MACCE - defined as the composite of death, Myocardial Infarction (MI), CerebroVascular Accident (CVA) or Stroke, or Target Vessel Revascularisation (TVR))

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Augustin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Mario C, Werner GS, Sianos G, Galassi AR, Buttner J, Dudek D, Chevalier B, Lefevre T, Schofer J, Koolen J, Sievert H, Reimers B, Fajadet J, Colombo A, Gershlick A, Serruys PW, Reifart N. European perspective in the recanalisation of Chronic Total Occlusions (CTO): consensus document from the EuroCTO Club. EuroIntervention. 2007 May;3(1):30-43. No abstract available. PMID 19737682
- [Background] Kahn JK. Angiographic suitability for catheter revascularization of total coronary occlusions in patients from a community hospital setting. Am Heart J. 1993 Sep;126(3 Pt 1):561-4. doi: 10.1016/0002-8703(93)90404-w. PMID 8362709
- [Background] Werner GS, Gitt AK, Zeymer U, Juenger C, Towae F, Wienbergen H, Senges J. Chronic total coronary occlusions in patients with stable angina pectoris: impact on therapy and outcome in present day clinical practice. Clin Res Cardiol. 2009 Jul;98(7):435-41. doi: 10.1007/s00392-009-0013-5. Epub 2009 Mar 18. PMID 19294443
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Garcia S, Sandoval Y, Roukoz H, Adabag S, Canoniero M, Yannopoulos D, Brilakis ES. Outcomes after complete versus incomplete revascularization of patients with multivessel coronary artery disease: a meta-analysis of 89,883 patients enrolled in randomized clinical trials and observational studies. J Am Coll Cardiol. 2013 Oct 15;62(16):1421-31. doi: 10.1016/j.jacc.2013.05.033. Epub 2013 Jun 7. PMID 23747787
- [Background] Sachdeva R. Effect of revascularization of chronic total occlusion on tandem stenoses in a "donor" artery. Tex Heart Inst J. 2014 Oct 1;41(5):547-50. doi: 10.14503/THIJ-13-3569. eCollection 2014 Oct. PMID 25425993
- [Background] Stone GW, Reifart NJ, Moussa I, Hoye A, Cox DA, Colombo A, Baim DS, Teirstein PS, Strauss BH, Selmon M, Mintz GS, Katoh O, Mitsudo K, Suzuki T, Tamai H, Grube E, Cannon LA, Kandzari DE, Reisman M, Schwartz RS, Bailey S, Dangas G, Mehran R, Abizaid A, Moses JW, Leon MB, Serruys PW. Percutaneous recanalization of chronically occluded coronary arteries: a consensus document: part II. Circulation. 2005 Oct 18;112(16):2530-7. doi: 10.1161/CIRCULATIONAHA.105.583716. No abstract available. PMID 16230504
- [Background] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612
- [Background] Olivari Z, Rubartelli P, Piscione F, Ettori F, Fontanelli A, Salemme L, Giachero C, Di Mario C, Gabrielli G, Spedicato L, Bedogni F; TOAST-GISE Investigators. Immediate results and one-year clinical outcome after percutaneous coronary interventions in chronic total occlusions: data from a multicenter, prospective, observational study (TOAST-GISE). J Am Coll Cardiol. 2003 May 21;41(10):1672-8. doi: 10.1016/s0735-1097(03)00312-7. PMID 12767645
- [Background] Srivatsa SS, Edwards WD, Boos CM, Grill DE, Sangiorgi GM, Garratt KN, Schwartz RS, Holmes DR Jr. Histologic correlates of angiographic chronic total coronary artery occlusions: influence of occlusion duration on neovascular channel patterns and intimal plaque composition. J Am Coll Cardiol. 1997 Apr;29(5):955-63. doi: 10.1016/s0735-1097(97)00035-1. PMID 9120181
- [Background] Katsuragawa M, Fujiwara H, Miyamae M, Sasayama S. Histologic studies in percutaneous transluminal coronary angioplasty for chronic total occlusion: comparison of tapering and abrupt types of occlusion and short and long occluded segments. J Am Coll Cardiol. 1993 Mar 1;21(3):604-11. doi: 10.1016/0735-1097(93)90091-e. PMID 8436741
- [Background] Rathore S, Matsuo H, Terashima M, Kinoshita Y, Kimura M, Tsuchikane E, Nasu K, Ehara M, Asakura Y, Katoh O, Suzuki T. Procedural and in-hospital outcomes after percutaneous coronary intervention for chronic total occlusions of coronary arteries 2002 to 2008: impact of novel guidewire techniques. JACC Cardiovasc Interv. 2009 Jun;2(6):489-97. doi: 10.1016/j.jcin.2009.04.008. PMID 19539251
- [Background] de Labriolle A, Bonello L, Roy P, Lemesle G, Steinberg DH, Xue Z, Kaneshige K, Suddath WO, Satler LF, Kent KM, Pichard AD, Lindsay J, Waksman R. Comparison of safety, efficacy, and outcome of successful versus unsuccessful percutaneous coronary intervention in "true" chronic total occlusions. Am J Cardiol. 2008 Nov 1;102(9):1175-81. doi: 10.1016/j.amjcard.2008.06.059. Epub 2008 Aug 27. PMID 18940287
- [Background] Suero JA, Marso SP, Jones PG, Laster SB, Huber KC, Giorgi LV, Johnson WL, Rutherford BD. Procedural outcomes and long-term survival among patients undergoing percutaneous coronary intervention of a chronic total occlusion in native coronary arteries: a 20-year experience. J Am Coll Cardiol. 2001 Aug;38(2):409-14. doi: 10.1016/s0735-1097(01)01349-3. PMID 11499731
- [Background] Hoye A, van Domburg RT, Sonnenschein K, Serruys PW. Percutaneous coronary intervention for chronic total occlusions: the Thoraxcenter experience 1992-2002. Eur Heart J. 2005 Dec;26(24):2630-6. doi: 10.1093/eurheartj/ehi498. Epub 2005 Sep 23. PMID 16183693
- [Background] Hannan EL, Racz M, Holmes DR, King SB 3rd, Walford G, Ambrose JA, Sharma S, Katz S, Clark LT, Jones RH. Impact of completeness of percutaneous coronary intervention revascularization on long-term outcomes in the stent era. Circulation. 2006 May 23;113(20):2406-12. doi: 10.1161/CIRCULATIONAHA.106.612267. Epub 2006 May 15. PMID 16702469
- [Background] Farooq V, Serruys PW, Garcia-Garcia HM, Zhang Y, Bourantas CV, Holmes DR, Mack M, Feldman T, Morice MC, Stahle E, James S, Colombo A, Diletti R, Papafaklis MI, de Vries T, Morel MA, van Es GA, Mohr FW, Dawkins KD, Kappetein AP, Sianos G, Boersma E. The negative impact of incomplete angiographic revascularization on clinical outcomes and its association with total occlusions: the SYNTAX (Synergy Between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery) trial. J Am Coll Cardiol. 2013 Jan 22;61(3):282-94. doi: 10.1016/j.jacc.2012.10.017. Epub 2012 Dec 19. PMID 23265332
- [Background] Patel VG, Brayton KM, Tamayo A, Mogabgab O, Michael TT, Lo N, Alomar M, Shorrock D, Cipher D, Abdullah S, Banerjee S, Brilakis ES. Angiographic success and procedural complications in patients undergoing percutaneous coronary chronic total occlusion interventions: a weighted meta-analysis of 18,061 patients from 65 studies. JACC Cardiovasc Interv. 2013 Feb;6(2):128-36. doi: 10.1016/j.jcin.2012.10.011. Epub 2013 Jan 23. PMID 23352817
- [Background] Prasad A, Rihal CS, Lennon RJ, Wiste HJ, Singh M, Holmes DR Jr. Trends in outcomes after percutaneous coronary intervention for chronic total occlusions: a 25-year experience from the Mayo Clinic. J Am Coll Cardiol. 2007 Apr 17;49(15):1611-1618. doi: 10.1016/j.jacc.2006.12.040. Epub 2007 Apr 2. PMID 17433951
- [Background] Christakopoulos GE, Christopoulos G, Carlino M, Jeroudi OM, Roesle M, Rangan BV, Abdullah S, Grodin J, Kumbhani DJ, Vo M, Luna M, Alaswad K, Karmpaliotis D, Rinfret S, Garcia S, Banerjee S, Brilakis ES. Meta-analysis of clinical outcomes of patients who underwent percutaneous coronary interventions for chronic total occlusions. Am J Cardiol. 2015 May 15;115(10):1367-75. doi: 10.1016/j.amjcard.2015.02.038. Epub 2015 Feb 18. PMID 25784515
- [Background] Tomasello SD, Boukhris M, Giubilato S, Marza F, Garbo R, Contegiacomo G, Marzocchi A, Niccoli G, Gagnor A, Varbella F, Desideri A, Rubartelli P, Cioppa A, Baralis G, Galassi AR. Management strategies in patients affected by chronic total occlusions: results from the Italian Registry of Chronic Total Occlusions. Eur Heart J. 2015 Dec 1;36(45):3189-98. doi: 10.1093/eurheartj/ehv450. Epub 2015 Sep 2. PMID 26333367
- [Background] Godino C, Bassanelli G, Economou FI, Takagi K, Ancona M, Galaverna S, Mangieri A, Magni V, Latib A, Chieffo A, Carlino M, Montorfano M, Cappelletti A, Margonato A, Colombo A. Predictors of cardiac death in patients with coronary chronic total occlusion not revascularized by PCI. Int J Cardiol. 2013 Sep 30;168(2):1402-9. doi: 10.1016/j.ijcard.2012.12.044. Epub 2013 Jan 12. PMID 23317549
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals (excerpts). J Am Coll Dent. 2014 Summer;81(3):23-30. PMID 25951680